CLINICAL TRIAL: NCT02264951
Title: Short Fatty Acids-induced Release of GLP-1 in Humans
Brief Title: Fat-induced Release of GLP-1 in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Katrine Bagge Hansen, MD, PhD, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SFAS
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Type 2 Diabetes
Keywords: Short fatty acids; 2-oleoyl glycerol; GLP-1 secretion; C8-diet oil; GIP secretion
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — tributyrin; Olive Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- A meal containing carrot and tributyrin (Active Comparator): A meal containing 200 g grated carrot and 0.0216 mol tributyrin; blood test taken from 0 - 2 hours postprandial
  Interventions: Dietary Supplement: Tributyrin; Dietary Supplement: Carrot
- A meal containing carrot and C8-diet oil (Active Comparator): A meal containing 200 g grated carrot and 0.0216 mol of C8-diet oil; blood test taken from 0 - 2 hours postprandial
  Interventions: Dietary Supplement: C8-diet oil; Dietary Supplement: Carrot
- A meal containing carrot and olive oil (Active Comparator): A meal containing 200 g grated carrot and 0.0216 mol of olive oil; blood test taken from 0 - 2 hours postprandial
  Interventions: Dietary Supplement: Olive oil; Dietary Supplement: Carrot
- A meal containing carrot (Placebo Comparator): A meal containing 200 g grated carrot; blood test taken from 0 - 2 hours postprandial
  Interventions: Dietary Supplement: Carrot

INTERVENTIONS:
Dietary Supplement: Tributyrin — a triglyceride containing three C4-acids
  Arms: A meal containing carrot and tributyrin
Dietary Supplement: C8-diet oil — a triglyceride containing 2 C8-fatty acids and one oleic acid at sn-2 position
  Arms: A meal containing carrot and C8-diet oil
Dietary Supplement: Olive oil — a triglyceride containing mostly three oleic acids
  Arms: A meal containing carrot and olive oil
Dietary Supplement: Carrot — mainly water and glucose

SUMMARY:
This study compared the incretin-releasing effect of C8-diet oil and tributyrin with that of 20 ml olive oil on a molar basis in human volunteers.

DETAILED DESCRIPTION:
A structured triglyceride (1,3-di-octanoyl-2-oleoyl-glycerol, called C8-diet oil), which upon digestion results in generation of two medium-chain fatty acids and 2-oleoyl-glycerol (2-OG), may lead to activation of GPR119 only, since medium fatty acids are poor agonists for fatty acid receptors.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian healthy male subjects
* Body mass index (BMI) 19 to 25 kg/m2
* Informed consent

Exclusion Criteria:

* Anaemia
* Diabetes mellitus
* Gastrointestinal diseases or operations interacting with intestinal absorption

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
plasma GLP-1 | 2 hours postprandial
plasma GIP | 2 hours postprandial

SECONDARY OUTCOMES:
plasma insulin | 2 hours postprandial
plasma PYY | 2 hours postprandial
plasma glucose | 2 hours postprandial
plasma neurotensin | 2 hour postprandial
plasma CCK | 2 hour postprandial

CONTACTS AND LOCATIONS:
Overall Officials: Jens J Holst, Professor, Study Chair — Biomedical Sciences, University of Copenhagen; Mette J Mandøe, Student, Principal Investigator — Glostrup Hospital; Biomedical Sciences, University of Copenhagen

REFERENCES:
- [Derived] Mandoe MJ, Hansen KB, Hartmann B, Rehfeld JF, Holst JJ, Hansen HS. The 2-monoacylglycerol moiety of dietary fat appears to be responsible for the fat-induced release of GLP-1 in humans. Am J Clin Nutr. 2015 Sep;102(3):548-55. doi: 10.3945/ajcn.115.106799. Epub 2015 Jul 15. PMID 26178726